CLINICAL TRIAL: NCT00612339
Title: Avastin in Combination With Temozolomide for Unresectable or Multifocal Glioblastoma Multiformes and Gliosarcomas
Brief Title: Avastin in Combination With Temozolomide for Unresectable or Multifocal GBMs and Gliosarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001022
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2012-09

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioma; Temozolomide; Temodar; Avastin; Bevacizumab; GBM; Gliosarcoma; Multifocal GBM; Brain tumor; Unresectable GBM; Glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin and Temozolomide (Experimental): Avastin administered at 10 mg/kg every 2 weeks beginning a minimum of 7 days after biopsy or 28 days after craniotomy. Temozolomide dosed at 200 mg/m2 daily for 5 days in a 28-day cycle.
  Interventions: Drug: Avastin and Temozolomide

INTERVENTIONS:
Drug: Avastin and Temozolomide — This is Phase II study with the combination of Avastin & Temozolomide for unresectable or multifocal WHO grade IV malignant glioma patients. Patients will receive up to 4 cycles of Avastin & Temozolomide . Avastin administered at 10 mg/kg every 14 days beginning minimum of 7 days after biopsy or 28 days after craniotomy. Temozolomide will be dosed at 200 mg/m2 daily x 5 days in 28-day cycle. Patients will have baseline MRI & repeat MRI every 4 weeks. If there is no evidence of disease progression after each cycle, or unacceptable toxicity, or as determined by investigators, patient non-compliance or patient withdraws consent to continue therapy & requests discontinuation, patients will receive up to 4 cycles of Avastin & Temozolomide, then proceed with standard XRT therapy, & future therapy after 4 cycles will be at discretion of patient & treating physicians.
  Other Names: Avastin - Bevacizumab; Temozolomide - Temodar

SUMMARY:
Primary objective- To determine efficacy of Avastin, 10 mg/kg every other week, in combination with standard 5-day temozolomide in terms of response rate.

Secondary objective- To determine safety of Avastin & Temozolomide in unresectable glioblastoma patients

DETAILED DESCRIPTION:
Subjects have histologically confirmed WHO gr IV primary malignant glioma that is unresectable/multifocal. This is Phase II study where up to 41 subjects will receive up to 4 cycles of Avastin & Temozolomide. Avastin administered at 10 mg/kg every 14 days beginning a minimum of 7 days after biopsy/28 days after craniotomy. Temozolomide dosed at 200 mg/m2 daily for 5 days in 28-day cycle. Patients will receive up to 4 cycles of Avastin & Temozolomide, then proceed with standard XRT. Study will use 2-stage "minimax" study design in which 21 subjects are accrued during 1st stage, with possibility that additional 20 patients accrued during 2nd stage. In initial Phase I & II trials, 4 potential Avastin-associated safety signals were identified: hypertension, proteinuria, thromboembolic events, & hemorrhage. Avastin-associated adverse events in Phase III trials include congestive heart failure, GI perforations, wound healing complications, & arterial thromboembolic events. Most common toxicity associated with Temozolomide has been mild myelosuppression.

ELIGIBILITY:
Inclusion Criteria:

Patients have histologically confirmed diagnosis of WHO gr IV primary malignant glioma. Patients will be unresectable or have multifocal disease.

* Age ≥ 18years & life expectancy of >12 weeks
* Evidence of measurable primary CNS neoplasm on contrast enhanced MRI.
* Interval of <1 week between prior biopsy/4 weeks from surgical resection & enrollment on protocol
* Karnofsky ≥60%
* Hemoglobin ≥9g/dl, ANC ≥1,500 cells/microliter, platelets ≥125,000 cells/microliter
* Serum creatinine ≤1.5 mg/dl, serum SGOT & bilirubin ≤1.5 x ULN
* For patients on corticosteroids, they must have been on stable dose for 1 week prior to entry, if clinically possible, & dose should not be escalated over entry dose level
* Signed informed consent approved by IRB prior to patient entry
* No evidence of > grade 1 CNS hemorrhage on baseline MRI/CT scan
* If sexually active, patients will take contraceptive measures for duration of treatments

Exclusion Criteria:

* Pregnancy/breast feeding
* Co-medication that may interfere with study results
* Active infection requiring IV antibiotics
* Prior or current Treatment w XRT/chemo for brain tumor, irrespective of grade of tumor
* Evidence of > grade 1 CNS hemorrhage on baseline MRI or CT scan

Avastin-Specific Concerns:

* Inadequately controlled hypertension
* Any prior history of hypertensive crisis/hypertensive encephalopathy
* New York Heart Association Grade II or > congestive heart failure
* History of myocardial infarction/unstable angina < 6 months prior to study enrollment
* History of stroke/transient ischemic attack < 6 months prior to study enrollment
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis/coagulopathy
* Major surgical procedure, open biopsy,/significant traumatic injury within 28 days prior to study enrollment/anticipation of need for major surgical procedure during course of study
* Core biopsy/other minor surgical procedure, excluding placement of vascular access device, <7 days prior to study enrollment
* History of abdominal fistula, GI perforation, /intra-abdominal abscess <6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either
* UPC ratio ≥1.0 at screening OR
* Urine dipstick for proteinuria ≥2+
* Known hypersensitivity to any component of Avastin
* Pregnant/lactating. Use of effective means of contraception in subjects of child-bearing potential
* Current, ongoing treatment with full-dose warfarin or its equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were accrued between October 2007 and September 2008 within the clinic at Duke Comprehensive Cancer Center.
Period: Overall Study
Arm/Group | Avastin and Temozolomide
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin and Temozolomide
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The proportion of subjects with complete or partial response as determined by a modification of the RANO (Response Assessment in Neuro-Oncology) criteria. A confirmation of response was not required. Complete Response was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks. Partial Response was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
Time Frame: 4 months
Population: All subjects
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Avastin and Temozolomide
Number analyzed (Participants) | 41
percentage of patients | 24.4 [12.4 to 40.3]

ADVERSE EVENTS:
Time Frame: 6 months
Description: CTCAE (3.0) was used for collecting adverse events in this study. However, the events have been converted to CTCAE (4.0) for entry into clinicaltrials.gov. Only grade 3, grade 4, and grade 5 adverse events were collected.
Arm/Group | Avastin and Temozolomide
Serious Adverse Events (participants affected / at risk) | 10/41
Other Adverse Events (participants affected / at risk) | 12/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin and Temozolomide (N=41)
ileus (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Death: Disease progression (General disorders) | 2
Anorectal infection (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin and Temozolomide (N=41)
Fatigue (General disorders) | 3
Platelet count decreased (Investigations) | 3
Peripheral motor neuropathy (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No